CLINICAL TRIAL: NCT03124472
Title: Effect of Uterine Artery Ligation Prior to Uterine Incision in Women With Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 169
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uterine artery ligation (Active Comparator): Pfannenstiel incision of skin and opening of the anterior abdominal wall in layers.
  * The loose peritoneum of the lower uterine segment is dissected downwards to mobilize the urinary bladder and expose the lower uterine segment.
  * Uterine artery ligation was performed by grasping the broad ligament with thumb anterior and the index finger lifting the base below the site uterine incision; the uterine artery was singly ligated with No. 1 vicryl suture. Myometrium was included so that uterine vessels are not damaged.
  * Cresenteric lower uterine segment incision was performed as usual. Higher incisions were performed in cases where the traditional incision was expected to be directly through the placenta.
  Interventions: Procedure: uterine artery ligation; Procedure: Lower segment Cesarean section
- Traditional lower segment Cesarean section (Active Comparator): Pfannenstiel incision of skin and opening of the anterior abdominal wall in layers.
  * The loose peritoneum of the lower uterine segment is dissected downwards to mobilize the urinary bladder and expose the lower uterine segment.
  * Cresenteric lower uterine segment incision was performed as usual. Higher incisions were performed in cases where the traditional incision was expected to be directly through the placenta.
  Interventions: Procedure: Lower segment Cesarean section

INTERVENTIONS:
Procedure: uterine artery ligation — Uterine artery ligation was performed by grasping the broad ligament with thumb anterior and the index finger lifting the base below the site uterine incision; the uterine artery was singly ligated with No. 1 vicryl suture. Myometrium was included so that uterine vessels are not damaged
  Arms: uterine artery ligation
Procedure: Lower segment Cesarean section — Pfannenstiel incision of skin and opening of the anterior abdominal wall in layers.
  - The loose peritoneum of the lower uterine segment is dissected downwards to mobilize the urinary bladder and expose the lower uterine segment.
  Cresenteric lower uterine segment incision was performed as usual. Higher incisions were performed in cases where the traditional incision was expected to be directly through the placenta Delivery of the baby and placenta.
  * Closure of the uterine incision in 2 layers with N0. 1 vicryl suture.
  * Closure of the anterior abdominal wall in layers

SUMMARY:
Pfannenstiel incision of skin and opening of the anterior abdominal wall in layers.

* The loose peritoneum of the lower uterine segment is dissected downwards to mobilize the urinary bladder and expose the lower uterine segment.
* Uterine artery ligation was performed by grasping the broad ligament with thumb anterior and the index finger lifting the base below the site uterine incision; the uterine artery was singly ligated with No. 1 vicryl suture. Myometrium was included so that uterine vessels are not damaged.
* Cresenteric lower uterine segment incision was performed as usual. Higher incisions were performed in cases where the traditional incision was expected to be directly through the placenta Delivery of the baby and placenta.
* Closure of the uterine incision in 2 layers with N0. 1 vicryl suture.
* Closure of the anterior abdominal wall in layers

DETAILED DESCRIPTION:
Pfannenstiel incision of skin and opening of the anterior abdominal wall in layers.

* The loose peritoneum of the lower uterine segment is dissected downwards to mobilize the urinary bladder and expose the lower uterine segment.
* Uterine artery ligation was performed by grasping the broad ligament with thumb anterior and the index finger lifting the base below the site uterine incision; the uterine artery was singly ligated with No. 1 vicryl suture. Myometrium was included so that uterine vessels are not damaged.
* Cresenteric lower uterine segment incision was performed as usual. Higher incisions were performed in cases where the traditional incision was expected to be directly through the placenta Delivery of the baby and placenta.
* Closure of the uterine incision in 2 layers with N0. 1 vicryl suture.
* Closure of the anterior abdominal wall in layers In the control group, lower segment caesarean section is without uterine artery ligation

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with placenta praevia antenatally
* plan is elective caesarean section
* Gestational age >34 weeks

Exclusion Criteria:

* Fetal distress
* medical disorders as hypertension or Diabetes Mellitus
* Coagulation defects.
* Emergency Cesarean section
* women with antepartum hemorrhage
* patients with marked ahdesions or those with non possible uterine artery ligation

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Decrease in Hemoglabin level | 24 hours after Cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes